CLINICAL TRIAL: NCT01177176
Title: Smoking Interventions for Hospital Patients: A Comparative Effectiveness Trial
Brief Title: Smoking Interventions for Hospital Patients
Acronym: Helping HAND
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Nancy A. Rigotti, Professor of Medicine, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1RC1HL099668 (NIH); 1RC1HL099668 (NIH)
Record Dates: First submitted 2010-08-03; First posted 2010-08-06 (Estimated); Last update posted 2014-09-18 (Estimated); Status verified 2014-09

CONDITIONS: Cigarette Smoking
Keywords: Cigarette smoking; Tobacco smoking
MeSH Terms: conditions — Cigarette Smoking; Tobacco Smoking | interventions — Nicotine Replacement Therapy; Bupropion; Varenicline; Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard Care (Other): Standard tobacco counseling provided to hospital inpatients as part of routine, clinical-guideline compliant care in the study hospital. No post-discharge treatment is offered in this arm.
  Interventions: Other: Standard Care
- Extended Care Management (Experimental): In addition to Standard Care, subjects in this arm receive Extended Care Management intervention to facilitate the continued use of smoking cessation treatment (counseling and medication use) after hospital discharge. This consists of 3 months of telephone-based contact after discharge.
  Interventions: Other: Extended Care Management

INTERVENTIONS:
Other: Extended Care Management — Telephone-based care management of tobacco cessation for 3 months after hospital discharge that features 2 innovations: (1) to increase medication use, smokers receive a free refillable 30-day sample of their choice of FDA-approved smoking cessation medication (nicotine replacement, bupropion, or varenicline) at hospital discharge; (2) to increase counseling cost-effectiveness, interactive voice recognition (IVR) technology is used to make automated telephone calls to identify the smokers seeking or most likely to benefit from continued counseling after hospital discharge.
  Other Names: nicotine replacement therapy; bupropion; varenicline; interactive voice response; telephone counseling for smoking cessation
  Arms: Extended Care Management
Other: Standard Care — Usual care provided to hospitalized smokers during their inpatient stay, with no post-discharge care management plan
  Arms: Standard Care

SUMMARY:
Cigarette smoking is the leading preventable cause of death in the U.S. Nearly 4 million U.S. smokers are hospitalized each year, many of them at high risk for tobacco-related disease or death. A hospital admission provides an opportunity for a smoker to quit. Smoking cessation counseling provided in the hospital is effective, but only if it continues for >1 month after discharge. Smoking cessation medications add benefit to counseling but are not often used. The challenge is to translate this efficacy research into routine clinical practice. The major barrier is to make the transition from inpatient to outpatient care. An evidence-based, cost-effective intervention model that can be adopted by U.S. hospitals is needed to realize the potential impact of hospital smoking interventions.

The Specific Aim of this project is to conduct a randomized controlled comparative effectiveness trial of two strategies to promote smoking cessation in hospitalized patients: (1) a hospital-only intervention that meets the current standard of the National Hospital Quality Measures("Standard Care"), and (2) an "Extended Care Management" model with 2 components that aims to encourage and facilitate the sustained use of smoking cessation treatment (counseling and medication use) after discharge in order to achieve long-term abstinence. It adds to Standard Care 3 months of telephone-based contact after discharge and feature 2 innovations: (1) to increase medication use, smokers willing to make a quit attempt receive a free, refillable 30-day sample of their choice of FDA-approved smoking cessation medication at hospital discharge; (2) to increase counseling cost-effectiveness, interactive voice recognition (IVR) technology is used to make automated telephone calls to identify the smokers interested in or most likely to benefit from continued counseling after discharge. The trial will enroll 330 adult smokers admitted to Massachusetts General Hospital, a 900-bed teaching hospital. Outcomes will be measured 1,3 and 6 months after hospital discharge. Study hypotheses are that the enhanced care arm, compared to usual care, is feasible and will increase (1) the use of smoking cessation treatment after discharge, (2) the duration of post-discharge tobacco abstinence, and (3) validated tobacco abstinence 6 months after hospital discharge (primary outcome). The principal secondary outcome measure is self-reported 7-day point prevalence tobacco abstinence after hospital discharge. Other secondary endpoints include self-reported point prevalence abstinence at 1 and 3 months, prolonged abstinence (self-reported tobacco abstinence at 1, 3, and 6 months). The cost-effectiveness (cost per quit) of the interventions will be also be compared.

ELIGIBILITY:
Inclusion Criteria:

* Cigarette smoker (daily smoker when smoking in usual way during the month before hospital admission)
* Counseled by hospital smoking counselor during hospital stay
* Plans to stop smoking tobacco products after hospital discharge
* Appropriate for use of smoking cessation medication after discharge

Exclusion Criteria:

* Expected hospital length of stay <24 hours
* Not expected to be discharged to home
* No access to a telephone
* Unable to communicate by telephone
* Severe psychiatric or neurologic disease precluding ability to be counseled
* Pregnant, nursing, or planning to become pregnant in next 3 months
* Active substance abuse other than tobacco
* Unable to speak English

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 397 (Actual)
Dates: Start 2010-07; Primary Completion 2012-11 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Validated 7-day point prevalence tobacco abstinence | 6 months after discharge
  7-day point prevalence tobacco abstinence, validated by saliva cotinine <= 10 ng/ml or if using NRT, expired air CO <=9ppm, or confirmation by proxy

SECONDARY OUTCOMES:
Use of tobacco treatment after hospital discharge | during 3 months and 6 months after hospital discharge
  patient-reported receipt of either smoking cessation counseling (defined as contact in person or by telephone) or smoking cessation pharmacotherapy (use of nicotine replacement therapy, bupropion, or varenicline)in the 3 months after hospital discharge
Duration of tobacco abstinence after hospital discharge | Up to 6 months after hospital discharge
  Number of days that patient reports not smoking any tobacco product after hospital discharge
Self-reported 7-day point prevalence tobacco abstinence | 6 month follow-up
Self-reported 7-day point prevalence tobacco abstinence | 3 months after hospital dicharge
Self-reported 7-day point prevalence tobacco abstinence | 1 month after hospital discharge
Prolonged tobacco abstinence | at 1, 3, and 6 months after hospital discharge
  Self-reported 7-day point prevalence abstinence at each of 3 time points: 1 month, 3 months, and 6 months after hospital discharge
Continuous tobacco abstinence | Up to 6 months after hospital discharge
  Self-reported continuous tobacco abstinence at (1) 1 month, (2) 3 months and (3) 6 months after hospital discharge

CONTACTS AND LOCATIONS:
Overall Officials: Nancy A Rigotti, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Result] Rigotti NA, Regan S, Levy DE, Japuntich S, Chang Y, Park ER, Viana JC, Kelley JH, Reyen M, Singer DE. Sustained care intervention and postdischarge smoking cessation among hospitalized adults: a randomized clinical trial. JAMA. 2014 Aug 20;312(7):719-28. doi: 10.1001/jama.2014.9237. PMID 25138333
- [Derived] Rigotti NA, Chang Y, Rosenfeld LC, Japuntich SJ, Park ER, Tindle HA, Levy DE, Reid ZZ, Streck J, Gomperts T, Kelley JHK, Singer DE. Interactive Voice Response Calls to Promote Smoking Cessation after Hospital Discharge: Pooled Analysis of Two Randomized Clinical Trials. J Gen Intern Med. 2017 Sep;32(9):1005-1013. doi: 10.1007/s11606-017-4085-z. Epub 2017 Jun 14. PMID 28616847
- [Derived] Duffy SA, Cummins SE, Fellows JL, Harrington KF, Kirby C, Rogers E, Scheuermann TS, Tindle HA, Waltje AH; Consortium of Hospitals Advancing Research on Tobacco (CHART). Fidelity monitoring across the seven studies in the Consortium of Hospitals Advancing Research on Tobacco (CHART). Tob Induc Dis. 2015 Sep 3;13(1):29. doi: 10.1186/s12971-015-0056-5. eCollection 2015. PMID 26336372
- [Derived] Japuntich SJ, Regan S, Viana J, Tymoszczuk J, Reyen M, Levy DE, Singer DE, Park ER, Chang Y, Rigotti NA. Comparative effectiveness of post-discharge interventions for hospitalized smokers: study protocol for a randomized controlled trial. Trials. 2012 Aug 1;13:124. doi: 10.1186/1745-6215-13-124. PMID 22852832